CLINICAL TRIAL: NCT04185142
Title: Combining Left Atrial Appendage Closure With Cryoballoon Ablation in Chinese Atrial Fibrillation Population
Brief Title: Combining Left Atrial Appendage Closure With Cryoballoon Ablation in Chinese Population
Acronym: CLACBAC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Ya-Wei Xu, Chief physician, Shanghai 10th People's Hospital
Other Study IDs: CLACBAC
Record Dates: First submitted 2019-11-25; First posted 2019-12-04 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: Atrial Fibrillation
Keywords: Combined procedure; Cryoballoon ablation; Left atrial appendage closure; Chinese
MeSH Terms: conditions — Atrial Fibrillation | interventions — Left Atrial Appendage Closure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- combined procedure group: patients underwent cryoballoon ablation and left atrial appendage closure
  Interventions: Combination Product: cryoballoon ablation combining with left atrial appendage closure

INTERVENTIONS:
Combination Product: cryoballoon ablation combining with left atrial appendage closure — cryoballoon ablation using either 1st or 2nd generation of cryoballoon and left atrial appendage closure using devices including WATCHMAN, Lefort and Lacbes.

SUMMARY:
Cryoablation combined with left atrial appendage closure is a novel strategy for atrial fibrillation patients. Through long-term follow-up, the investigators aimed to observe the safety and efficacy of the combined procedure in Chinese population.

DETAILED DESCRIPTION:
the investigators aimed to observe the clinical outcome of combining cryoballoon ablation (CBA) with left atrial appendage closure (LAAC) in drug-refractory non-valvular atrial fibrillation patients, who have high risk of stroke or hemorrhage, or contraindication of long-term oral anticoagulants (OACs).

The combined procedure was completed using CBA following LAAC. Generally, 3-month OACs, following 3-month double antiplatelet therapy, and lifelong single platelet therapy was recommended as antithrombotic regimen.

At 3rd,6th,12th and every year after since the procedure, Holter and transoesophageal echocardiography monitoring, and outpatient follow-up was applied to every patient.

The safety was evaluated by all-cause mortality, peri- and postprocedural complications. While the efficacy was evaluated through the freedom of atrial arrhythmia, stroke incidence, and withdrawal of OACs.

ELIGIBILITY:
Drug refractory non-valvular paroxysmal atrial fibrillation patients,

Inclusion Criteria:

1. CHA2DS2-VASc score≥2 or HAS-BLED score≥3,
2. having contraindications to long-term oral anticoagulants (OACs),
3. refuse OAC therapy despite explanation.

Exclusion Criteria:

1. thrombus in left atrium (LA) or left atrial appendage (LAA) presented and confirmed by transoesophageal echocardiograph (TEE),
2. oversized LA (LA diameter>65mm by TTE) or LAA (LAA opening>35mm) through TEE,
3. pericardial effusion (≥4mm by TTE or TEE),
4. hemodynamic unstable patients,
5. patients with active hemorrhagic diseases,
6. ischemic or hemorrhagic stroke within 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chinese with documented non-valvular atrial fibrillation who meet the inclusion criteria while without any of the exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2015-10-16 (Actual); Primary Completion 2023-11-16 (Estimated); Study Completion 2024-11-16 (Estimated)

PRIMARY OUTCOMES:
Recurrence of atrial arrhythmia | since the start of the procedure, third, sixth, twelfth month, and every year after, up to 5 years.
  The proportion of patients have recurrent atrial arrhythmia, including atrial tachycardia lasting longer than 30 seconds, atrial flutter, and atrial fibrillation. Detected by either ECG or 24 Holter monitor.
Incidence of stroke | since the start of the procedure, third, sixth, twelfth month, and every year after, up to 5 years.
  the proportion of patients have either hemorrhagic or ischemic stroke confirmed by CT or MRI.

SECONDARY OUTCOMES:
All-cause death | since the start of the procedure, third, sixth, twelfth month, and every year after, up to 5 years.
  Death event due to any cause
Cardiovascular death | since the start of the procedure, third, sixth, twelfth month, and every year after, up to 5 years.
  death due to cardiovascular cause
Major hemorrhagic events | since the start of the procedure, third, sixth, twelfth month, and every year after, up to 5 years.
  Intracranial hemorrhage, gastrointestinal bleeding, or any overt bleeding with hemoglobin drop ≥3 to 5 g/dL.
Myocardial infarction | since the start of the procedure, third, sixth, twelfth month, and every year after, up to 5 years.
  Diagnosed myocardial infarction with or without ST segment elevation.
Peripheral vascular embolism | since the start of the procedure, third, sixth, twelfth month, and every year after, up to 5 years.
  Arterial or venous thrombosis except cardiac or cerebral vascular embolism confirmed by imaging examination.
Rehospitalization due to cardiovascular events | Since the start of the procedure to 5 years.
  Inpatient admission or emergency department admission with cardiovascular causes.
Redo-ablation | since the start of the procedure, third, sixth, twelfth month, and every year after, up to 5 years.
  Ablation intended to treat recurrent atrial arrhythmia
Withdrawal of oral anticoagulants | since the start of the procedure, third, sixth, twelfth month, and every year after, up to 5 years.
  The proportion of patients stop oral anticoagulation therapy including warfarin, dabigatran, or rivaroxaban.
Residual flow | Instantly after the procedure, and the 3rd month after the procedure. Evaluation at 1 year will be arranged according to the last TEE result.
  Residual flow between LAAC device and LAA measured by TEE
LAAC device position | Instantly after the procedure, and the 3rd month after the procedure. Evaluation at 1 year will be arranged according to the last TEE result.
  displacement of LAAC device evaluated by TEE
Device related thrombus | Instantly after the procedure, and the 3rd month after the procedure. Evaluation at 1 year will be arranged according to the last TEE result.
  Thrombus surrounding or attached to the LAAC device detected by TEE
Atrioesophageal fistula | Instantly after the procedure, and the 3rd month after the procedure. Evaluation at 1 year will be arranged according to the last TEE result.
  Fistula between left atrium and esophagus detected by TEE.
Pericardial effusion | Since the start of the procedure, third, sixth, twelfth month, and every year after, up to 5 years.
  Any amount of pericardial effusion detected by TTE or TEE

CONTACTS AND LOCATIONS:
Overall Officials: Yawei Xu, MD, PhD, Principal Investigator — Department of Cardiology, Shanghai Tenth People's Hospital
Locations (1):
- Department of Cardiology, Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Ren Z, Zheng Y, Zhang J, Yang H, Wu J, Li H, Guo R, Meng W, Zhang J, Sun H, Xu Y, Zhao D. Patients With Larger Left Atrial Appendage Orifice Presented Worse Prognosis Contributed by Acute Heart Failure After Left Atrial Appendage Closure. J Am Heart Assoc. 2022 Sep 20;11(18):e026309. doi: 10.1161/JAHA.122.026309. Epub 2022 Sep 14. PMID 36102232